CLINICAL TRIAL: NCT03540628
Title: A Single Center, Investigator Blinded, Randomized Placebo Control, 24 Month, Parallel Group, Superiority Study to Compare the Efficacy of Thiamine, Vitamin C and Hydrocortisone in the Treatment of Septic Shock.
Brief Title: Thiamine, Vitamin C and Hydrocortisone in the Treatment of Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health South (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MMMC#1576
Record Dates: First submitted 2018-02-26; First posted 2018-05-30 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Thiamine; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Enrollment for this study will be initiated in patients with septic shock that require addition of a second pressor agent.
  The control arm of our randomized trial will receive a second pressor agent, hydrocortisone and standard of care. If the patient needs additional pressor support or therapy, that will be recorded in the results.
  The experimental arm will receive a second pressor agent and hydrocortisone, plus thiamine and vitamin C along with the standard of care. If the patient needs additional pressor support or therapy that will be recorded in the results.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Eligible patients will be randomized in equal blinded proportions by the pharmacy department to receive thiamine, vitamin C and hydrocortisone in the experimental arm or continue with hydrocortisone plus placebo and usual standard of care treatment as discussed previously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Arm (No Intervention): The control arm of our randomized trial will receive a second pressor agent, hydrocortisone and standard of care to care for septic shock. The IV bags will be blinded by pharmacy. If the patient needs additional pressor support or therapy, the data will be recorded in the results.
- Thiamine and Vitamin C administration Arm (Experimental): The experimental arm will receive a second pressor agent and hydrocortisone, plus thiamine and vitamin C along with the standard of care. The IV bags will be blinded by pharmacy. If the patient needs additional pressor support or therapy, the data will be recorded in the results.
  Interventions: Dietary Supplement: Thiamine and Vitamin C

INTERVENTIONS:
Dietary Supplement: Thiamine and Vitamin C — Supplementary vitamins for the patient in septic shock
  Arms: Thiamine and Vitamin C administration Arm

SUMMARY:
The purpose of this research study is to determine whether patients who receive thiamine (vitamin B1), vitamin C and hydrocortisone while in septic shock have improved outcomes compared to hydrocortisone alone.

A recently published article "Hydrocortisone, Vitamin C and Thiamine for the treatment of Severe Sepsis and Septic Shock," suggested substantial mortality reduction (78%). We wish to test the hypothesis that mortality reduction is at least 25% in a prospective randomized trial. Other important sub-aims include the testing whether the protocol reduces the time on pressors agents, reduces the trajectory of the SOFA score, or reduces the trajectory of procalcitonin.

DETAILED DESCRIPTION:
The study has four specific aims. The first is to utilize the Marik protocol published in CHEST to determine mortality reduction in septic shock with thiamine (vitamin B1), vitamin C and hydrocortisone supplementation. The second aim is to determine whether supplementation with thiamine, vitamin C and hydrocortisone reduce time spent on vasopressor support. Thirdly, whether the trajectory of the SOFA score is affected by supplementation with thiamine, hydrocortisone and vitamin C. Fourthly, assess the trajectory of procalcitonin, a laboratory test, in patients treated with the protocol.

This is a single center community based hospital in Southwest Michigan, investigator blinded, randomized placebo controlled trial, 24 month, parallel group, two arm, superiority study with a 1:1 allocation ratio to compare the efficacy of thiamine, vitamin C and hydrocortisone in the treatment of severe sepsis and septic shock. Each arm of the research study will contain 30 patients in order to detect a 25% mortality reduction. Enrollment for this study will be initiated in patients with septic shock that require addition of a second pressor agent. The control arm of our randomized trial will receive a second pressor agent, hydrocortisone and standard of care. If the patient needs additional pressor support or therapy, that will be recorded in the results.

The experimental arm will receive a second pressor agent and hydrocortisone, plus thiamine and vitamin C along with the standard of care. If the patient needs additional pressor support or therapy that will be recorded in the results.

To clarify, both arms will utilize two vasopressor agents, hydrocortisone and supportive care, the experimental group will also receive vitamin C and thiamine.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Septic Shock on two vasopressor agents
2. Age between 18-90 years old
3. Ability to provide written informed consent

Exclusion criteria include:

1. Age younger than 18 years old
2. Pregnancy
3. DNR or DNI status with limitations of care, such as "supportive care only"
4. Patients/advocates that request thiamine, vitamin C or hydrocortisone supplementation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The mortality rate comparison of patients with septic shock at Lakeland Regional Medical Center to the study published in CHEST. | 24 months
  The mortality rate difference between control and experimental arms

SECONDARY OUTCOMES:
The duration on vasopressor support | 24 months
  Control and Experimental arms will quantify the time requiring vasopressor therapy.
Quantify the Sequential Organ Failure Assessment score in Septic shock patients requiring vasopressor therapy | 24 months
  Control and experimental arms with both calculate daily Sequential Organ Failure Assessment scores to assess for differences.

CONTACTS AND LOCATIONS:
Locations (1):
- Lakeland Regional Healthcare, Saint Joseph, Michigan, United States

IPD SHARING:
Plan to Share IPD: No